CLINICAL TRIAL: NCT03845686
Title: Brain Markers Predicting Reading Recovery After Stroke
Status: Completed | Type: Observational
Sponsor: Kessler Foundation (Other)
Collaborators: Rutgers University (Other); National Center for Medical Rehabilitation Research (NCMRR) (NIH)
Responsible Party: Principal Investigator, Olga Boukrina, Research Scientist, Kessler Foundation
Other Study IDs: R-784-13
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-04

CONDITIONS: Left-Hemisphere Stroke
Keywords: stroke; reading; fMRI; perfusion; activation; BOLD; recovery; subacute; chronic
MeSH Terms: conditions — Stroke; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subacute Stroke Sample: Participants with first-ever left-brain stroke, < 4 weeks post stroke, age >18 years, right-handed, fluent and literate in English prior to stroke, no prior neurological disorders or clinical stroke event, <4 weeks post-stroke; able to undergo an MRI and complete study tasks, and presence of reading deficits.
  Interventions: Diagnostic Test: Perfusion functional Magnetic Resonance Imaging (perfusion fMRI)
- Chronic Stroke Sample: The same group of participants examined in the chronic post-stroke period (>3 months post-stroke)
  Interventions: Diagnostic Test: Perfusion functional Magnetic Resonance Imaging (perfusion fMRI)

INTERVENTIONS:
Diagnostic Test: Perfusion functional Magnetic Resonance Imaging (perfusion fMRI) — The goal of this test is to measure brain activity during subacute and chronic post-stroke period using a widely available non-invasive neuroimaging tool - functional Magnetic Resonance Imaging (fMRI). Because fMRI relies in part on cerebral blood flow, which is altered in stroke, measuring longitudinal changes in neural activity with fMRI requires that we control for concomitant changes in blood circulation. To do this, we will employ a novel dual-echo perfusion fMRI sequence, which will allow us to separately estimate neural and vascular contributions to fMRI.

SUMMARY:
For millions of stroke survivors acquired reading deficits represent a significant handicap preventing them from returning to work or continuing their education. The goal of the proposed research is to investigate what brain mechanisms enable recovery of impaired reading. To achieve this goal, the project will directly measure changes in brain perfusion (blood flow) and activation among recovering stroke survivors using a neuroimaging technique called perfusion fMRI (functional Magnetic Resonance Imaging). The project will test if re-perfusion (return of circulation) and re-appearance of reading-related brain activity in the left-brain network for reading is associated with recovery. The ability to predict recovery from neuroimaging has tremendous value in rehabilitation for generating prognoses. It may also dramatically improve the quality of research evaluation for novel, targeted interventions such as noninvasive brain stimulation or pharmacologic therapies.

DETAILED DESCRIPTION:
There is a fundamental gap in understanding the neuro-behavioral time-course of reading recovery following stroke. It is not known whether recovery of reading is associated with improved blood circulation and neural activity of the peri-infarct area, or whether circulation in the unaffected, contralateral brain areas contributes to functional recovery. Continued existence of this gap represents an important problem because, until it is filled, knowledge about optimal timing and targets for restorative therapies to improve reading will remain out of reach. The long-term goal is to develop clinical prognostic and therapeutic tools to improve reading limitations. The overall objective of this project is to characterize the neural mechanisms of recovery from stroke-induced reading impairments. The central hypothesis of this study is that subacute-to-chronic recovery of reading ability is potentiated by reperfusion (improved blood flow) of the left reading network. Reperfusion promotes the return of neural activity and supports behavioral recovery. In contrast, increased perfusion of the right brain areas represents a maladaptive response and is associated with worse chronic reading ability. This hypothesis has been formulated on the basis of preliminary data. The rationale for the proposed research is that once the neural recovery from stroke-induced reading impairments is characterized, clinicians will be able to predict individual recovery potential and select appropriate rehabilitation goals. Guided by strong preliminary data, this hypothesis will be tested by pursuing two specific aims: 1) Determine whether post-stroke changes in cerebral blood flow predict recovery of reading ability; and 2) Determine whether increased baseline perfusion of the left reading network is paralleled by greater reading-related neural activation. Under the first aim, perfusion in the peri-infarct tissue, left reading network, and homologous right brain areas will be examined among left stroke patients with reading impairments. A non-invasive measure of perfusion (Arterial Spin Labeling, ASL MRI) will be applied longitudinally: <4 weeks post-stroke (sub-acute) and >3 months post-stroke (chronic) to test if increased perfusion of the left reading network is coupled with an improvement of reading accuracy. Under the second aim, reading-induced brain activity will be recorded in the same group of patients using perfusion-based functional MRI. The effect of task-related neural activity on recovery will be separated from the effect of cerebral blood flow by statistically controlling for baseline circulation and by modeling independent contributions of perfusion and BOLD (Blood Oxygen Level Dependent) signals in order to estimate cerebral oxygen consumption rate, which is directly related to neural activity. The conceptual innovation of this study is that it offers the opportunity to examine reading recovery as distinct from other functions. The methodological innovation is in using simultaneously-acquired perfusion and BOLD signals, helping to measure longitudinal changes in circulation and neural activity with unprecedented precision. The proposed research is significant because it can help greatly improve the effectiveness of post-stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* right-handed
* fluent and literate in English prior to stroke
* no prior neurological disorders or clinical stroke event
* <4 weeks post-stroke
* ability to undergo an MRI and complete study tasks
* presence of reading deficits

Exclusion Criteria:

* participants with severe aphasia resulting in severe language deficits and inability to consent
* participants with very large lesions resulting in severe cognitive deficits and inability to consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 34 participants with first-ever left-brain stroke
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Reading Aloud Accuracy - subacute | within 1 week of study enrollment
  Percent correct of single words read aloud
Reading Aloud Accuracy - chronic | 3 months after study enrollment
  Percent correct of single words read aloud
Phonology Task Accuracy - subacute | within 1 week of enrollment
  2-alternative forced choice task of pseudoword rhyming
Phonology Task Accuracy - chronic | 3 months after study enrollment
  2-alternative forced choice task of pseudoword rhyming
Semantics Task Accuracy - subacute | within 1 week of enrollment
  2-alternative forced choice task of picture matching
Semantics Task Accuracy - chronic | 3 months after study enrollment
  2-alternative forced choice task of picture matching
Orthography Task Accuracy - subacute | within 1 week of enrollment
  2 alternative forced choice between a correctly spelled word and a phonological foil
Orthography Task Accuracy - chronic | 3 months after study enrollment
  2 alternative forced choice between a correctly spelled word and a phonological foil
Perfusion MRI - subacute | within 1 week of enrollment
  Subacute cerebral blood flow (CBF) in peri-infarct tissue, left reading network, and right homologous areas
Perfusion MRI - chronic | 3 months after enrollment
  Subacute-to-chronic change of CBF in peri-infarct tissue, left reading network, and right homologous areas
Functional MRI - subacute | within 1 week of enrollment
  Brain activation for reading words and nonwords; task-induced change in oxygen consumption
Functional MRI - chronic | 3 months after enrollment
  Subacute-to-chronic change of brain activation for reading words and pseudowords; longitudinal and task-induced change in oxygen consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated in this project may be shared in accordance with the NIH and Kessler Foundation policies, as well as the Notice of Privacy of Practices signed by each participant in the study. In case data is shared, it will be de-identified, such that no link can be made to the individual participant. Data may be shared upon request after the acceptance for publication of the main findings of the study. Publication of findings will occur during the project, if appropriate, or at the conclusion of the project, consistently with the typical scientific process.
  Access to methodology and software tools generated in the course of the project will be granted for educational, research, and non-profit purposes. Sharing of such study resources will be provided via web-based applications (e.g., GitHub), as appropriate.
Time Frame: The data will be available 1 year after study completion (3/31/2021 - anticipated). The data will be available indefinitely
Access Criteria: The data will be made available upon request